CLINICAL TRIAL: NCT03711955
Title: The Improvement in Cognitive and Motor Function: An 8 Week Study Comparing the Effects of Instability Resistance Training Versus Aerobic Training on Cognitive and Motor Improvements Found in Parkinson's Disease Participants.
Brief Title: Comparing the Effects of Instability Resistance Training Versus Aerobic Training on Cognitive and Motor Improvements Found in Parkinson's Disease Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Alisha Mistry, Primary Investigator, Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Sunlife1
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Exercise; Parkinson Disease
MeSH Terms: conditions — Motor Activity; Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the aerobic training group/intervention or the instability resistance training group/intervention
Who Masked: Participant, Investigator
Masking Description: Investigator will not engage in the 8 week training program occurring, a leading supervisor will lead every training session so that the primary investigator (myself) will be blinded to the participants and their performance throughout the 8 week training interventions.
  Participants from the opposite training groups will have separate training session times. In this way, no participant from the opposite training group will have contact with each other (ex. aerobic training group's session is at 12pm; instability resistance training group's session is at 4pm).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training group (AET) (Experimental): Each AET sessions are to last one hour, with 40 minutes being allocated to the aerobic exercise training component, 10 minutes allocated to warm-ups, 5 minutes allocated to cool-downs, and one 5 minute rest period between the 20 minutes spent on each machine (20 minutes of cycling, 5 minute rest, 20 minutes seated row). The AET program consists of 20 minutes of cycling on the stationary bicycle and 20 minutes of seated row on the kinesis Technogym machine. This is to be preceded by 10 minutes of static stretching during warm up, and 5 minutes of post-exercise recovery (dynamic stretches).
  Interventions: Other: Exercise
- Instability training group (IRT) (Experimental): Each IRT sessions are to last one hour, with time being allocated to a 10 minute warm up, consisting of static stretches, a 5 minute cool down, consisting of dynamic stretches, and a series of IRT exercises performed in a circuit setting over the duration of 40 minutes. In the sessions, five resistance exercises will be performed. A linear periodization will occur, in which the training load will progress from high-volume low-intensity to low-volume high-intensity loads over the duration of eight weeks to maximize training adaptations. Additionally, there will be a progressive increase in load/resistance by 1-2 lbs and the degree of instability of each exercise during the course of the eight week program. Unstable devices will be changed from the least unstable to the most unstable device throughout the program, but only when participants showed a considerable decrease in body sway/movement and force production increased when performing exercises.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Two types of training exercises, AET and IRT, will be used as the interventions in this study. Participants will either be assigned to the AET group or the IRT group, where they will participate in the respective training intervention group for 8 consecutive weeks.

SUMMARY:
This study will be looking at the effects that instability resistance training and aerobic training, individually, have on the improvement of various motor and cognitive impairments present in individuals with Parkinson' disease.

There will be 25-30 participants in this study (all of whom have Parkinson's disease). Once passing the eligibility criteria, participants will complete as series of baseline/pre-tests and then be randomly assigned to either the aerobic training group or the instability training group, where they will participate in every training session that occurs in the next 8 consecutive weeks. There will be 3 training sessions a week occurring on non-consecutive days (ex. Monday, Wednesday, Friday) for both training groups (3 aerobic training sessions, 3 instability resistance training sessions). Once the 8 week training intervention has been completed, a series of post-tests will occur exactly once week after (same tests used as in the pre-tests)

DETAILED DESCRIPTION:
Twenty-eight to thirty selected participants that fit the eligibility criteria will go through a series of baseline (pre-test) tests during screening session. It should be noted that all participants are to be assessed in their clinical "ON" state (fully medicated).Motor and cognitive tests are conducted to determine the baseline level of participants in the following domain of motor and cognitive functions:

1. Timed Up and Go test: mobility test measuring participants static and dynamic balance on gait mat (Protokinetic gait mat)
2. Protokinetic gait mat: measure gait velocity and spatial and temporal gait variability (stride length, stride time, double support time, and step width)

   a.Measured through three tests: i.dual-tasking walking (counting backwards from 15, naming countries) ii.walking at normal speed (3 trails) iii.fast walking
3. Grip Strength test: measure overall strength
4. Unified Parkinson's Disease Rating Scale (UPDRS): assess various motor, cognitive, emotional and activities of daily living components of Parkinson's disease
5. Montreal Cognitive Assessment (MoCa) test: assess cognitive domains and look for Mild Cognitive Impairment (MCI) (attention and concentration, executive functions, memory, language) with scores ranging from 13-24
6. Trail-Making Test: tests visual attention and task-switching Part A: includes number 1-25, must draw lines and connect numbers in ascending order Part B: includes both letters and numbers; must draw lines connecting number and letters in ascending order ( but must alternate between number and letters, ex. 1-A-2-B)
7. Delis-Kaplan Executive Function System: executive function deficits, those being: measurement of selective attention and cognitive flexibility Trial 1: participant would say out loud the patches of colour Trial 2: participant would read words out loud printed in black ink Trial 3: participant has to say the ink colour, not the word Trial 4: participant has to say the ink colour, not the word UNLESS the word is in a box, then the participant has to say the word and not say the ink colour.
8. Parkinson Disease Cognitive Rating Scale : comprehensive cognitive function scale (measuring frontal sub-cortical and posterior cortical tasks)

Intervention Once baseline tests are completed, participants will be randomly assigned into either the instability resistance training group or the aerobic training group (done through RANDOM.org database), with each group receiving equal number of participants. Participants will participate in an eight week training program that will begin within one week after the baseline tests are completed. This training program will run over the course of eight weeks, with scheduled training sessions occurring three times a week (Monday, Wednesday, Friday), and will be running for one hour for both AET and IRT training groups. In total, there will be a total of twenty-four training sessions for both AET and IRT groups.

Aerobic Training

Each AET sessions are to last one hour, with 40 minutes being allocated to the aerobic exercise training component, 10 minutes allocated to warm-ups, 5 minutes allocated to cool-downs, and one 5 minute rest period between the 20 minutes spent on each machine (ex. 20 minutes of cycling, 5 minute rest, 20 minutes seated row). The AET program consists of 20 minutes of cycling on the stationary bicycle and 20 minutes of seated row on the kinesis Techno-gym machine. This is to be preceded by 10 minutes of static stretching during warm up, and 5 minutes of post-exercise recovery (dynamic stretches). The exercise intensity on both modalities (rowing machine and recumbent bicycle) is to be maintained throughout sessions by using the following checklist: 1) maintaining 70% of maximum heart rate (HRmax) predicted by age (determined by the formula HRmax=208-(0.7× age), 2) maintaining a pace of 50rpm, and 3) maintain a score below 5 on the Borg rating 10-point scale. Additionally, the resistance are to be kept at a constant weight throughout the 20 minutes of cycling and seated row, and is to only be increased/decreased when 1) participants are below the 70% maximum heart rate (HRmax) and/or 2) participants have a score above 5 on the Bohr scale (in which resistance/weights will be decreased). Each session will be led by lab supervisors/coordinators along with trained volunteers. The supervisors and volunteers will demonstrate, guide, monitor and assists participants in the exercises if required.

Instability Resistance Training

Each IRT sessions are to last one hour, with time being allocated to a 10 minute warm up, consisting of static stretches, a 5 minute cool down, consisting of dynamic stretches, and a series of IRT exercises performed in a circuit setting over the duration of 40 minutes. Just as the AET sessions, IRT sessions will run for one hour, three times a week, for eight-weeks. Before the beginning of the first session, a baseline performance is to be completed for every participant, to determine their 1 repetition maximum (RM) on each exercise modality. Once the baseline tests are completed, participants will begin their exercise sessions. In the sessions, five resistance exercises will be performed (reverse lunge row, half squats, ankle plantar flexion, push-ups, and trunk rotations). All the exercises shown, except push-ups, will be performed on the Techno-gym Kinesis machine. A linear periodization will occur, in which the training load will progress from high-volume low-intensity to low-volume high-intensity loads over the duration of eight weeks to maximize training adaptations(number of sets increase and the number of repetitions decrease). Additionally, there will be a progressive increase in load/resistance by 1-2 lbs and the degree of instability of each exercise during the course of the eight week program. Unstable devices will be changed from the least unstable to the most unstable device throughout the program (balance pad, balance discs, dyna discs, Swiss ball, BOSU ball), but only when participants showed a considerable decrease in body sway/movement and force production increased when performing exercises (ability to balance body on device and maintain center of mass). Furthermore, these devices are placed between the base of support for each participant and the floor. If participants are not able to perform an exercise with higher loads/resistance due to the increase in instability of new unstable device, participants must maintain the same load used in previous session. Rest time will be allocated throughout each session (30sec-1min rests between each set). Each session will be monitored, guided and assisted by leading lab supervisor/coordinator along with trained volunteers. The supervisors and volunteers will demonstrate, guide, monitor and assists participants in the exercises if required.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease participants aged between 50 to 80 years old
* Has idiopathic Parkinson's disease
* On stable medication (dopaminergic medication)
* Hoehn and Yahr stage between 2 and 3
* Does not present other neurological disorder other than Parkinson's disease)
* Does not have significant arthritis, cardiovascular disease, and cognitive impairment by Mini-Mental State Examination (score <23)
* Has normal or corrected vision in at one eye in order to carry out exercise)
* Able to comply to scheduled visits, treatments, and other trial procedures
* Must be in sufficient health to participate in study's training program as determined through the use of Physical Activity Readiness Questionnaire-Plus (PARQ+) screening tool, coupled with evaluation by a certified exercise physiologist/physician for clearance to participate in training program

Exclusion Criteria:

* has uncontrolled hypertension and/or diabetes
* Is currently participating in any form of physical activity/exercise program that involves AET or RT two or more times a week in the last six months
* presence of dementia which is determined by having a score of 13 or less on the MoCa test.
* has significant arthritis, cardiovascular disease, and cognitive impairment by Mini-Mental State Examination (score <23)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
executive function (memory, language and concentration) | change from baseline executive functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  memory, language and concentration will be measured using Montreal Cognitive Assessment test
executive function (selective attention, cognitive flexibility) | change from baseline executive functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  selective attention, cognitive flexibility will be measured using the Delis-Kaplan Executive Function System test
executive function (visual attention and task switching) | change from baseline executive functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  visual attention and task switching ability will be measured using the Trail Making Test
executive function (attention, working memory and recall verbal memory) | change from baseline executive functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  sustained attention, working memory, and immediate and delayed free recall verbal memory is measured using the Parkinson's Disease Cognitive Rating Scale (score total out of 134-the perfect score. The closer to 134, the the better results)
gait variability | change from baseline gait functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  gait variability will be measured using the the Protokinetic Gait-walk test
muscular strength | change from baseline muscular strength tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  muscular strength will be measured using the grip strength test (jamar dynamometer tool)
gait (static and dynamic balance) | change from baseline gait functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  static and dynamic balance will be measured using Timed Up and Go Test
assessing comprehensive motor and non-motor symptoms | change from baseline motor and non-motor functions tested after 8 weeks of intervention (post-test measured on consecutive week after last week of intervention)
  assess non-motor experiences of daily living, motor experiences of daily living, motor examination, and motor complications symptoms will be assessed through the Unified Parkinson's Disease Rating Scale (0-4 rating scale, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Alisha Mistry, Principal Investigator — Movement Disorder Research and Rehabilitation Center
Locations (1):
- Movement Disorder Research and Rehabilitation Centre, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: synergic trail — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-018-0782-7
- See also: balance and fear of falling in subjects with Parkinson's disease is improved after exercises with motor complexities — https://www.ncbi.nlm.nih.gov/pubmed/29310015
- See also: resistance training with instability for patients with Parkinson's disease — https://www.ncbi.nlm.nih.gov/pubmed/27054681
- See also: symptom and gait changes after sensory attention focused exercise vs aerobic training in Parkinson's disease — https://www.ncbi.nlm.nih.gov/pubmed/19373930